CLINICAL TRIAL: NCT06123624
Title: Comparison of Desflurane and Sevoflurane on Remifentanil Requirement Using Analgesia Nociception Index-guided Anesthesia
Brief Title: Desflurane and Sevoflurane on Remifentanil Requirement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJOUIRB-IV-2023-380
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane group (Experimental)
  Interventions: Drug: Desflurane Inhalation Solution
- Sevoflurane group (Placebo Comparator)
  Interventions: Drug: Sevoflurane Inhalation Solution

INTERVENTIONS:
Drug: Desflurane Inhalation Solution — Keeping the anesthesia using desflurane inhalation solution as 1 minimal alveolar concentration
  Arms: Desflurane group
Drug: Sevoflurane Inhalation Solution — Keeping the anesthesia using sevoflurane inhalation solution as 1 minimal alveolar concentration
  Arms: Sevoflurane group

SUMMARY:
The primary purpose of this study is to compare the desflurane and sevoflurane on remifentanil requirement using analgesia nociception index-guided anesthesia in patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of herniated disc, injury of spinal cord, and neoplasm of spinal meninges

Exclusion Criteria:

* Hyperbilirubinemia
* Prior chronic pain
* Prior opioid abuse
* Cardiac arrythmia

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
remifentanil requirement | at time of the end of skin suture (up to 3 hours)
  assessing the total dose of remifentanil administered from skin incision until skin suture